CLINICAL TRIAL: NCT01787630
Title: Initiating Phase II-III Study to Evaluate the Technique and Effects of Separating the Prostate From the Rectum With Hyaluronic Acid During Radiotherapy
Brief Title: To Evaluate the Technique and Effects of Separating the Prostate and Rectum With Hyaluronic Acid During Radiotherapy
Acronym: NoHarm
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anders Widmark (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Sponsor-Investigator, Anders Widmark, Professor, MD, Umeå University
Organization: Umeå University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NoHarm1
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Prostatic Cancer
Keywords: Prostatic cancer; Radiotherapy; Hyaluronic acid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronic acid (Experimental): Hyaluronic acid will be injected in the space between the prostate and rectum prior to radiotherapy to perform a dorsal movement of rectum.
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Device: Hyaluronic acid — Injection in connection with ultrasound
  Other Names: NASHA Spacer Gel

SUMMARY:
The dominating problem after local radiotherapy of prostate cancer is rectal toxicity. If the rectum could be completely moved out of the treated volume, a substantial decrease of rectal toxicity seems reasonable. In this study we will develop and evaluate a new transrectal injection technique where hyaluronic acid (HA) is injected in the space between the prostate and the rectum prior to external beam radiotherapy to increase the physical distance between prostate and rectum.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified prostatic cancer
* Low or intermediate risk prostatic cancer
* Lymph node negative
* Suitable for radiotherapy

Exclusion Criteria:

* Earlier treatment for prostatic cancer
* Unable to co-operate or suffering from any other form of disease that would interfere with the planned treatment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-01; Primary Completion 2016-03 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Remaining volume of HA | 24 month after end of radiotherapy
  Measurement on the remaining volume of HA by MRI

SECONDARY OUTCOMES:
Quality of life | 24 month after end of radiotherapy
  Patient evaluation with questionnaires regarding Quality of Life and side effects after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Anders Widmark, Prof MD, Principal Investigator — Umea university, dept of oncology
Locations (3):
- Sweden (3):
  - Department of oncology, Kalmar Hospital, Kalmar
  - Department of oncilogy, Sundsvall Hospital, Sundsvall
  - Department of oncology, University Hospital, Umeå